CLINICAL TRIAL: NCT02794974
Title: Ultrasound-guided Intermediate Cervical Plexus Block for Carotid Endarterectomies
Brief Title: Ultrasound-guided Intermediate Cervical Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Research Center (Other)
Responsible Party: Principal Investigator, Dr.med.Ronald Seidel, MD, Helios Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 2016-0027
Record Dates: First submitted 2016-05-31; First posted 2016-06-09 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Internal Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Cervical Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with perivascular block (Experimental): 1. ultrasound-guided intermediate cervical plexus block (20ml ropivacaine 0.75%) 2. facial nerve block (cervical branch) (5ml prilocaine 1%) 3. perivascular block (5ml prilocaine 1%)
  Interventions: Other: cervical plexus block; Other: facial nerve block; Other: perivascular block
- without perivascular block (Experimental): 1. ultrasound-guided intermediate cervical plexus block (20ml ropivacaine 0.75%) 2. facial nerve block (cervical branch) (5ml prilocaine 1%)
  Interventions: Other: cervical plexus block; Other: facial nerve block

INTERVENTIONS:
Other: cervical plexus block — ultrasound-guided application of 20ml ropivacaine 0.75%
  Other Names: cervical plexus anesthesia
Other: facial nerve block — ultrasound-guided application of 5ml prilocaine 1%
  Other Names: facial nerve anesthesia
Other: perivascular block — ultrasound-guided application of 5ml prilocaine 1%
  Other Names: perivascular infiltration
  Arms: with perivascular block

SUMMARY:
The investigators test with the present study design, whether an ultrasound-guided blockade of the cervical plexus in combination with an additional application of local anesthetic to the superficial cervical ansa (facial nerve: cervical branch) leads to an improved quality of anesthesia.

DETAILED DESCRIPTION:
The innervation of the neck area is complex and includes cranial nerve (innervation of the vessel wall (IX,X) and of the neck muscles (VII,XI)), as well as the cervical plexus and brachial plexus. This is a major cause of insufficient anesthesia quality during carotid endarterectomies.

The investigators test with the present prospective study design, whether an ultrasound-guided blockade of the cervical plexus in combination with an additional application of local anesthetic to the superficial cervical ansa (facial nerve: cervical branch) leads to an improved quality of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* internal carotid stenosis: open surgical revascularization
* age over 18 years
* written informed consent

Exclusion Criteria:

* allergy (local anesthetics)
* pregnancy
* participation in other studies
* drug addiction
* non-cooperative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Seidel, MD, Principal Investigator — Helios Medical Center Schwerin, Department of Anesthesiology and Intensive care,
Locations (1):
- Helios Medical Center Schwerin, Department of Anaesthesiology and Intensive Care, Schwerin, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited as part of the preoperative information discussion. All patients received an intermediate cervical plexus block and a facial nerve block (cervical branch, superficial cervical ansa). The decision on an additional perivascular infiltration was made by an experienced physician on the basis of sonoanatomic properties.
Groups:
- Cervical Plexus and Facial Nerve Block: 1. ultrasound-guided intermediate cervical plexus block (20ml ropivacaine 0.75%) 2. block of the facial nerve (cervical branch) (5ml prilocaine 1%)
  cervical plexus block: ultrasound-guided application of 20ml ropivacaine 0.75%
  facial nerve block: ultrasound-guided application of 5ml prilocaine 1%
- Cervical Plexus, Perivascular and Facial Nerve Block: 1. ultrasound-guided intermediate cervical plexus block (20ml ropivacaine 0.75%) 2. block of the facial nerve (cervical branch) (5ml prilocaine 1%) 3. perivascular local anesthetic infiltration (5ml prilocaine 1%)
  cervical plexus block: ultrasound-guided application of 20ml ropivacaine 0.75%
  facial nerve block: ultrasound-guided application of 5ml prilocaine 1%
  perivascular block: ultrasound-guided application of 5ml prilocaine 1%
Period: Overall Study
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Started | 14 | 15
Completed | 14 | 14
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Plexus, Perivascular and Facial Nerve Block | Cervical Plexus and Facial Nerve Block | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9) | 71 (10) | 69 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 8 | 13 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Local Anesthetic Supplementation (Frequency)
Description: number of participants who need supplementation of prilocaine 1% by the surgeon (%)
Time Frame: intraoperatively
Measure: Number; unit: participants
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Number analyzed (Participants) | 14 | 14
participants | 11 | 7
Statistical Analysis 1: Comparison: Cervical Plexus and Facial Nerve Block vs Cervical Plexus, Perivascular and Facial Nerve Block; Test type: Superiority; p = 0.236, Fisher Exact

2. Primary Outcome: Local Anesthetic Supplementation (Volume)
Description: volume of prilocaine 1% supplemented by the surgeon (ml)
Time Frame: intraoperatively
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Number analyzed (Participants) | 14 | 14
ml | 4.2 (3.1) | 1.7 (2.0)
Statistical Analysis 1: Comparison: Cervical Plexus and Facial Nerve Block vs Cervical Plexus, Perivascular and Facial Nerve Block; Test type: Superiority; p = 0.018, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Hoarseness
Description: number of participants who experienced side effects: hoarseness
Time Frame: intraoperatively
Measure: Number; unit: participants
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Number analyzed (Participants) | 14 | 14
participants | 8 | 12
Statistical Analysis 1: Comparison: Cervical Plexus and Facial Nerve Block vs Cervical Plexus, Perivascular and Facial Nerve Block; Test type: Superiority; p = 0.209, Odds Ratio; Odds Ratio = 4.5, 95% CI 2-sided [0.63 to 32.2]

4. Secondary Outcome: Cough
Description: number of participants who experienced side effects: cough
Time Frame: intraoperatively
Measure: Number; unit: participants
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Number analyzed (Participants) | 14 | 14
participants | 4 | 7
Statistical Analysis 1: Comparison: Cervical Plexus and Facial Nerve Block vs Cervical Plexus, Perivascular and Facial Nerve Block; Test type: Superiority; p = 0.44, Odds Ratio; Odds Ratio = 2.5, 95% CI 2-sided [0.49 to 12.77]

5. Secondary Outcome: Dysphagia
Description: number of participants who experienced side effects: dysphagia
Time Frame: intraoperatively
Measure: Number; unit: participants
Arm/Group | Cervical Plexus and Facial Nerve Block | Cervical Plexus, Perivascular and Facial Nerve Block
Number analyzed (Participants) | 14 | 14
participants | 4 | 6
Statistical Analysis 1: Comparison: Cervical Plexus and Facial Nerve Block vs Cervical Plexus, Perivascular and Facial Nerve Block; Test type: Superiority; p = 0.695, Odds Ratio; Odds Ratio = 1.88, 95% CI 2-sided [0.37 to 9.45]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Without Perivascular Block | With Perivascular Block
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02794974/SAP_001.pdf
  • Study Protocol (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT02794974/Prot_002.pdf